CLINICAL TRIAL: NCT02977624
Title: Effectiveness of a Telerehabilitation Intervention to Improve Activity and Participation Among Adults Following Acquired Brain Injury
Brief Title: A Telerehabilitation Intervention to Improve Activity and Participation Among Adults Following Acquired Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0689-15-HMO
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Brain Injury, Chronic
MeSH Terms: conditions — Brain Injury, Chronic

STUDY DESIGN:
Intervention Model Description: This exploratory study was a partially randomized controlled trial with a waitlist control crossover design.

ARMS (2):
- Tele-CO-OP (Experimental): The intervention included weekly videoconferencing sessions using the Cognitive Orientation to Daily Occupational Performance approach (tele-CO-OP) over a period of three months. Participant identified five functional goals, of which three were directly addressed.
  Interventions: Behavioral: The Cognitive Orientation to daily Occupational Performance
- Waitlist control (No Intervention): The waitlist control group did not receive the intervention during the same time period

INTERVENTIONS:
Behavioral: The Cognitive Orientation to daily Occupational Performance
  Arms: Tele-CO-OP

SUMMARY:
Objectives - To evaluate the effectiveness of an telerehabilitation intervention program among acquired brain injury (ABI) survivors in the chronic phase. The aim of the intervention is to improve the transition from rehabilitation units to community dwelling and facilitate activity and participation in life roles in the community.

Working hypothesis - The telerehabilitation based program for ABI survivors will be effective in:

1. Improving function in activities of daily living, participation in occupations and health related quality of life.
2. Reducing the need for outpatient clinic and rehabilitation services.
3. The intervention achievements will be maintained in 3-month follow-up

Methodology - Participants: ABI survivors will be selected from patients who are referred to the outpatient or home-based rehabilitation unit of Maccabi health services. Following completion of out-patient occupational therapy treatment in the rehabilitation centers the participants will be randomly assigned into two groups: The treatment group will receive the intervention program in addition to standard care, and the waitlist control group will receive standard care only.

Outcome measures:

1. The Canadian Occupational Performance Measure (COPM)
2. The Performance Quality Rating Scale (PQRS)
3. Mayo-Portland Adaptability Inventory (MPAI-4)
4. The Dysexecutive Questionnaire (DEX)
5. The New General Self-Efficacy Scale (NGSE)
6. The Zarit Caregiver Burden Scale short version

Procedure: The intervention program includes up to 20 video sessions over 3 months between an occupational therapist and the participant. The virtual meetings will be conducted using The Cognitive Orientation to daily Occupational Performance approach. The meetings will focus on problem solving for daily life situations and on the ability to implement the discussed strategies for a variety of activities. Participants will be evaluated at baseline, after the intervention, and after 6 months.

DETAILED DESCRIPTION:
The intervention program includes up to 20 video sessions over 3 months between an occupational therapist and the participant. The virtual meetings will be conducted using The Cognitive Orientation to daily Occupational Performance approach. The meetings will focus on problem solving for daily life situations and on the ability to implement the discussed strategies for a variety of activities. Participants will be evaluated at baseline, after the intervention, and after 6 months.

ELIGIBILITY:
Inclusion Criteria:

(1) ≥ 6 months post-ABI; (2) age ≥ 18 years; (3) sufficient proficiency in Hebrew or English to participate in the study; (4) modified Rankin scale (mRS) scores of 2-4 reflecting slight to moderate disability [38]; (5) self-reported unmet functional goals; (6) internet access at home; and (7) had an adult significant other who agreed to be involved in the study

Exclusion Criteria:

(1) moderate or severe aphasia; (2) a score of <21 on the Mini Mental Status Examination (MMSE) or Montreal Cognitive Assessment scores: MOCA<19; (3) dementia diagnosis; (3) an acute illness which significantly impacts the ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
The Canadian Occupational Performance Measure (COPM) | 6 months: baseline, post intervention (after 3 months), follow-up (after 3 more months)
  The COPM is a semi-structured interview to facilitate client-centered goal setting and measure the client's perceived occupational performance and satisfaction levels.
The Performance Quality Rating Scale (PQRS) | 6 months: baseline, post intervention (after 3 months), follow-up (after 3 more months)
  The PQRS is an observational measure of activity performance.
The Mayo-Portland Adaptability Inventory (MPAI-4) | 6 months: baseline, post intervention (after 3 months), follow-up (after 3 more months)
  The MPAI-4 measures the recovery progress of people after an ABI and includes 29 items grouped into three subscales: (a) Ability (e.g., motor, sensory and cognitive abilities), (b) Adaptation (e.g., emotional state and social interactions), and (c) Participation (e.g., leisure activities, employment and transportation).

SECONDARY OUTCOMES:
The Dysexecutive Questionnaire (DEX) | 6 months: baseline, post intervention (after 3 months), follow-up (after 3 more months)
  The DEX is a 20-item questionnaire to assess executive function in daily life among people with ABI
The New General Self-Efficacy Scale (NGSE) | 6 months: baseline, post intervention (after 3 months), follow-up (after 3 more months)
  This is an 8-item questionnaire that assesses people's confidence in their ability to accomplish their goals, regardless of the obstacles they may face
the Short Form Zarit Burden Interview | 6 months: baseline, post intervention (after 3 months), follow-up (after 3 more months)
  A measure of caregiver burden

OTHER OUTCOMES:
Satisfaction questionnaire | Post intervention
  A measure of the participants' satisfaction with the tele-CO-OP intervention
Background questionnaire | 6 months: baseline, post intervention (after 3 months), follow-up (after 3 more months)
  A questionnaire to document sociodemographic and clinical characteristics